CLINICAL TRIAL: NCT07278076
Title: Clinical Decision-Making During FEES: The Impact of Residue Amount and Location
Acronym: IRAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25093017
Record Dates: First submitted 2025-11-17; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Decision Making
Keywords: clinical decision making; pharyngeal residue severity interpretation
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Thirty (50%) of the clinicians participating in the study will watch a 30-minute educational presentation about current research on clinical decision making and aspiration risks of pharyngeal residue after the image assessment task is completed. Several peer-reviewed articles will be presented via video recording. These articles support several key tenets of this research study. These clinicians would then re-test. Using this information, the PI will compare diet restriction patterns between the education (treatment) and no-education (control) groups, potentially demonstrating whether knowledge dissemination can reduce fear-based decision-making. Ordinal logistic regression will be used to examine if any significance difference between the control and experimental groups exists. Any identified significant differences could help change how FEES is conducted and interpreted.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Identifying the threshold for allowed residue amount and location (No Intervention): The first aim of this study is to identify the threshold of the volume and location of residue at which clinicians restrict diets. In the quantitative study, clinicians will be presented with the same case study. In the case study, the patient participates in a FEES and two randomized images at a time are displayed to the clinician to represent the patient's valleculae and pyriform sinuses. Each image of the set will have varying amounts of residue. The amount of residue will be controlled to represent each level of pharyngeal residue (i.e. none, trace, mild, moderate, and severe) according to the standardized and validated Yale Pharyngeal Residue Severity Rating. Each participant will score 25 combinations of location and severity. Using a five-point Likert scale, the participants will rate how likely they are to restrict the patient's diet based on the amount of pharyngeal residue displayed in both the valleculae and pyriform sinuses.
- Educational intervention is provided (Experimental): Thirty (50%) of the clinicians participating in the study will watch a 30-minute educational presentation about current research on clinical decision making and aspiration risks of pharyngeal residue after they complete the image assessment task (Specific Aim 1). Several peer-reviewed articles will be presented via video recording. These clinicians would then re-test. Using this information, the PI will compare diet restriction patterns between the education (treatment) and no-education (control) groups, potentially demonstrating whether knowledge dissemination can reduce fear-based decision-making. Ordinal logistic regression will be used to examine if any significance difference between the control and experimental groups exists. Any identified significant differences could help change how FEES is conducted and interpreted.
  Interventions: Other: education
- Clinician interview during the qualitative portion of this study (No Intervention): The third aim of this study is to explore the rationale behind the clinician's decision-making. Participants from the quantitative portion of this mixed-methods study will be prompted to justify their clinical reasoning in the second part of the study, during an interview. Independent interviews will be conducted to reduce clinician influences. This aim should help identify possible fear-based decision-making by the clinicians when assessing amounts of pharyngeal residue. The questions presented will also serve to understand if or how clinicians follow evidence-based guidelines during FEES. A semi-structured format will be utilized to allow for follow-up questions. In collecting data, a descriptive approach will be used that is bottom up. A phenomenological inquiry will be utilized to investigate the thought process of each clinician as they navigate through the various factors that can impact their decision to restrict a diet consistently.

INTERVENTIONS:
Other: education — In the second aim of the study, 30 (50%) of the clinicians participating in the study will watch a 30-minute educational presentation about current research on clinical decision making and aspiration risks of pharyngeal residue after they complete the image assessment task (Specific Aim 1). Several peer-reviewed articles will be presented via video recording. These articles support several key tenets of this research study and include: 1) recommendations should be based on clinical experience and training, not evidence-based practice,8 2) the location of pharyngeal residue does not increase or decrease penetration or aspiration risk,6 and 3) a correlation, not a causation exists between the amount of pharyngeal residue and aspiration risk.14 Other studies indicated that other factors should be investigated, such as the accumulation of residue over time.14 These clinicians would then re-test.
  Arms: Educational intervention is provided

SUMMARY:
In this study, the investigator aims to identify the threshold of food residue visualized in the throat during a FEES (fiberoptic endoscopic evaluation of swallowing) that speech-language pathologists allow before restricting a patient from eating. 60 speech-language pathologists will be required to participate, with half of them watching a pre-recorded video detailing current research about residue in the throat of pharynx. The group watching the video will then re-score their images. This investigates the impact of education on clinical decision-making. Finally, 8 clinicians will meet with the researcher individually to share their clinical decision-making rationale. With this information, the researcher hopes to identify a patient population who is at risk for diet restrictions in order to encourage speech-language pathologists to extend the swallow study and trial more compensatory strategies before restricting the patient's diet.

DETAILED DESCRIPTION:
The purpose of this research is to identify the location and threshold of pharyngeal residue at which clinicians restrict diets for patients in the outpatient setting. 60 clinicians will judge 25 pairs of photos from FEES (fiberoptic endoscopic evaluation of swallowing) where each of the five levels of pharyngeal residue (e.g. none, trace, mild, moderate, and severe) are represented. These levels are used by the standardized and validated Yale Pharyngeal Residue Severity Rating Scale (YPRSRS).11 Residue severity in both the valleculae and pyriform sinuses will be presented, creating 25 image combinations. The patient history for each pair of photographs is the same: no airway compromise has occurred, the patient is ambulatory, does not require supplemental oxygen, has no cognitive deficits and is receiving out-patient care. Clinicians will indicate at which severity level of pharyngeal residue they are most likely to restrict the diet using a Likert scale (e.g. "extremely unlikely", "unlikely", "neutral", "likely", and "extremely unlikely"). Observing diet restrictions when pharyngeal residue reaches moderate levels would support our hypothesis that clinicians make risk-averse recommendations.

The other aim of this project is to evaluate the impact of evidence-based education on clinician decision-making regarding pharyngeal residue and location. Half of the clinicians will be randomized to the treatment group and watch a recorded 30-minute pre-recorded video presentation about research on pharyngeal residue before they complete the image assessment task. Using this information, a comparison can be made with diet restriction patterns between the educated (treatment) and non-educated (control) groups, potentially demonstrating whether evidence-based clinical research reduces fear-based decision-making. Should the investigators observe that the experimental group restricts diets less than the control group, the hypothesis that clinicians and patients benefit from evidence-based clinical education would be accurate.

Finally, the researcher would like to determine the rationale behind clinician decision-making. During the qualitative portion of this study, the researcher will interview eight clinicians. Clinicians will be chosen from the original group of 60 to participate in a structured interview to investigate the rationale behind their clinical decision-making. An analysis will be completed to determine the distribution of clinicians who chose to restrict the diet compared to those who did not. The clinicians chosen will reflect the ratio of restrictive and non-restrictive clinicians. The researchers anticipate that clinicians who watched the recorded research presentation are less likely to restrict diets based on pharyngeal residue alone regardless of the location. In collecting data, a bottom-up descriptive approach will be utilized. A phenomenological framework will investigate the various factors that might impact a clinician's decision to restrict a diet.

ELIGIBILITY:
Inclusion Criteria:

* Speech language pathologists with at least one year of experience conducting FEES (flexible endoscopic evaluations of swallowing)

Exclusion Criteria:

* Anyone who is not a speech pathologist, or has less than one year of experience conducting FEES.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
If a diet restriction occurs based on the residue amount and location | In one year since the initiation of the study
  Clinicians will be rating if they would restrict an oral diet based on pictures of pharyngeal residue of various amounts (none, trace, mild, medium, severe) in two locations: the valleculae and pyriform sinuses.

SECONDARY OUTCOMES:
Identifying if education impacts how pharyngeal residue is interpreted | In one year since the initiation of the study
  The secondary measure is to identify if education (a pre-recorded presentation on up to date dysphagia management research) impacts how clinicians interpret the amount and location of pharyngeal residue during FEES. Clinicians will first rate randomized photos of pharyngeal residue of each category. Then the clinicians will watch a video, and will have to re-rate randomized photos. The amounts of pharyngeal residue will be categorized as none, trace, mild, moderate and severe based on the Yale Pharyngeal Residue Severity Rating Scale. Pictures presented will show each residue amount in two locations; the pyriform sinuses and valleculae. Clinicians will indicate if they would restrict oral eating based on the picture of pharyngeal residue.
Ivestigating the rationale behind clinical decision making during pharyngeal residue management | In one year since the initiation of the study
  8 clinicians will be chosen to be interviewed to investigate the rationale behind their clinical decision-making